CLINICAL TRIAL: NCT06269562
Title: Postoperative Analgesic Efficacy of Clavipectoral Plan Block and Serratus Posterior Superior Intercostal Plane Block Combination in Clavicle Surgeries: A Report of Five Cases
Brief Title: SPSIPB and CPB on Clavicle Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Fatih Balci, Specialist Doctor, Department of Anesthesiology and Reanimation, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: clavicle
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Clavicle Fracture; Postoperative Pain; Analgesia
Keywords: serratus posterior superior intercostal plane block; clavipectoral plane block; clavicle fracture; pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Block (Experimental): consists of 5 patients in whom both techniques were applied
  Interventions: Procedure: Serratus posterior superior intercostal plane block and clavipectoral plane block

INTERVENTIONS:
Procedure: Serratus posterior superior intercostal plane block and clavipectoral plane block — The analgesic effectiveness achieved by the concurrent application of these two techniques was investigated.

SUMMARY:
Clavicular fractures represent a common occurrence often necessitating effective pain management strategies, particularly following surgical interventions. This study involved a cohort of five patients who underwent clavicular fracture surgery under general anesthesia. A novel analgesic approach combining two distinct nerve block techniques-Serratus Posterior Superior Intercostal Plane Block (SPSIPB) and Clavipectoral Plane Block (CPB)-was employed for postoperative pain control. The procedural methodology encompassed the administration of SPSIPB preceding anesthesia induction, followed by CPB subsequent to induction. SPSIPB targeted specific neural regions responsible for sensory blockade within the innervation of the clavicular skin, whereas CPB focused on the clavipectoral fascia. Standard anesthesia protocols were utilized, and postoperative pain levels were evaluated using Numeric Rating Scores (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Five American Society of Anesthesiologists (ASA) Ⅰ-II- III patients scheduled for clavicle surgery will be included in the study

Exclusion Criteria:

* patients with bleeding disorders
* patients with signs of infection in the block application area
* patients with unstable haemodynamics
* patients with thyroid cardiovascular, renal, hepatic and neuropsychiatric diseases
* patients with vascular disease,
* patients with respiratory distress
* patients whose consent for the study could not be obtained or who did not accept to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 24 hours after the procedure
  0=no pain , 10= the worst pain

SECONDARY OUTCOMES:
tramadol consumption | 24 hours after the procedure
  total tramadol consumption of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No